CLINICAL TRIAL: NCT07328893
Title: Effect of Single Dose Intravenous Magnesium Sulfate on Postoperative Analgesic Consumption in Patients Undergoing Laparoscopic Cholecystectomy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tata Main Hospital (Other)
Responsible Party: Principal Investigator, Dr.Deb Sanjay Nag, Chief Consultant & HOD, Tata Main Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TP250122626
Record Dates: First submitted 2025-12-27; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Analgesia; Postoperative
MeSH Terms: conditions — Agnosia | interventions — Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Intervention Model Description: The central research question revolves around whether a single intravenous dose of magnesium sulfate can effectively reduce postoperative analgesic consumption in this patient population.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Triple-blind: not only from participants and administrators, but also from those tasked with analyzing the data after the experiment has concluded. Masking will be done by independent caregivers making the drug or the palcebo (drug) in look alike syringes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MgSO4(Group: M) (Experimental): The Magnesium Sulfate Group (M), receiving 30 mg/kg intravenous magnesium sulfate diluted in 100 ml Normal Saline at the induction of anesthesia,
  Interventions: Drug: Magnesium Sulfate 30 mg/kg intravenous diluted in 100 ml Normal Saline.
- Normal Saline (Group: S) (Placebo Comparator): The Placebo Group Group (S) will recieve 100 ml Normal Saline at the induction of anesthesia.
  Interventions: Drug: Magnesium Sulfate 30 mg/kg intravenous diluted in 100 ml Normal Saline.

INTERVENTIONS:
Drug: Magnesium Sulfate 30 mg/kg intravenous diluted in 100 ml Normal Saline. — Patients will be randomly assigned to one of two groups: the Magnesium Sulfate Group (M), receiving 30 mg/kg intravenous magnesium sulfate diluted in 100 ml Normal Saline at the induction of anesthesia, or the Normal Saline Group (S), receiving an equivalent volume of Normal Saline. Both groups will also receive standard multimodal analgesia with intravenous Diclofenac (75 mg) and Paracetamol (1 gm) at the time of port closure.

SUMMARY:
This study describes a randomized controlled trial designed to evaluate the impact of a single intravenous dose of magnesium sulfate on postoperative analgesic consumption in patients undergoing laparoscopic cholecystectomy. The primary aim is to determine if magnesium sulfate can reduce postoperative morphine usage and its associated side effects.

The study will involve 106 patients (53 per arm), aged 18-65, classified as ASA physical status I or II, who are scheduled for elective laparoscopic cholecystectomy. Participants will be randomly assigned to receive either 30 mg/kg intravenous magnesium sulfate or a placebo (normal saline), alongside standard anesthetic care. Secondary outcomes include pain scores, the time until rescue analgesia is needed, and the monitoring of hemodynamic responses and potential adverse events. Statistical analysis will utilize descriptive statistics, chi-square tests, and t-tests or Mann-Whitney U-tests to compare the two groups.

DETAILED DESCRIPTION:
This study describes a meticulous randomized controlled trial designed to investigate the "Effect of single dose intravenous magnesium sulfate on postoperative analgesic consumption in patients undergoing laparoscopic cholecystectomy." The study addresses a critical clinical need, as laparoscopic cholecystectomy, despite being a minimally invasive procedure, often leads to significant postoperative pain. This pain traditionally necessitates opioid analgesics, which, while effective, come with a host of undesirable side effects such as nausea, vomiting, constipation, dizziness, and even respiratory depression. The study aims to explore multimodal analgesia (MMA) by specifically examining magnesium, a known NMDA receptor antagonist with analgesic properties, as a means to reduce opioid dependency and improve patient recovery.

The central research question revolves around whether a single intravenous dose of magnesium sulfate can effectively reduce postoperative analgesic consumption in this patient population. The null hypothesis posits that intravenous magnesium sulfate will decrease analgesic consumption, while the alternate hypothesis suggests no such effect.

The primary objective is to quantify the reduction in postoperative morphine consumption in the magnesium group compared to the placebo. Secondary objectives are comprehensive, including the evaluation of pain intensity using the Visual Analogue Scale (VAS), the time until patients require rescue analgesia, an assessment of hemodynamic stability, the impact on neuromuscular blockade, and the incidence of any other adverse events.

Methodologically, it will be a parallel, two-arm randomized controlled trial. Eligible participants will be adult patients (18-65 years) classified as ASA Physical status I or II, scheduled for elective laparoscopic cholecystectomy. Stringent exclusion criteria are in place to ensure patient safety and data integrity, covering factors like patient refusal, high BMI, obstructive sleep apnea, significant organ dysfunction, certain medication use, substance abuse, psychiatric illness, specific surgical durations, or conversion to open surgery.

Patients will be randomly assigned to one of two groups: the Magnesium Sulfate Group (M), receiving 30 mg/kg intravenous magnesium sulfate diluted in 100 ml Normal Saline at the induction of anesthesia, or the Normal Saline Group (S), receiving an equivalent volume of Normal Saline. Both groups will also receive standard multimodal analgesia with intravenous Diclofenac (75 mg) and Paracetamol (1 gm) at the time of port closure. Rescue analgesia, in the form of Morphine (3-4 mg), will be administered if a patient's VAS score is ≥ 4. Extensive intraoperative and postoperative monitoring will be conducted to track various physiological parameters and pain-related outcomes. A robust sample size of 117 patients (53 per arm, adjusted for a 10% attrition rate) has been determined to ensure sufficient statistical power (90%) to detect a 30% reduction in morphine use, with a two-sided significance level of 5%. Data analysis will be performed using SPSS, employing descriptive statistics, Chi-square tests for categorical variables, and independent samples t-tests or Mann Whitney U-tests for continuous variables, with a P-value < 0.05 considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

Age - 18 - 65 years, either sex American Society of Anesthesiologists (ASA) Physical status classification system group I and II Elective laparoscopic cholecystectomy

Exclusion Criteria:

Patient refusal BMI > 30 kg/m² OSA Renal, hepatic or cardiovascular dysfunction including cardiac conduction disorders Those on long term calcium channel blockers or receiving magnesium supplements Opioid or analgesic abuse Psychiatric illness Surgical duration < 1 h & > 3 h Lap converted to open

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-12-27 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Total dose of post-operative morphine consumption. | 24 hours
  Rescue analgesia, in the form of Morphine (3-4 mg), will be administered if a patient's VAS score is ≥ 4.

SECONDARY OUTCOMES:
Post operative Pain Scores Pain | 24 hours
  Visual Analogue Scale
Time to rescue analgesic | 24 hours
  Time after the surgery when the patient asks for rescue analgesic or the patient's VAS score is ≥ 4.

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - Tata Main Hospital, Jamshedpur, Jharkhand
  - Dr.Deb Sanjay Nag, Jamshedpur, Jharkhand

IPD SHARING:
Plan to Share IPD: No
Can be shared as per GDPR guidelines masking individual patient details.